CLINICAL TRIAL: NCT00519987
Title: An Open Label, Single Center Study to Assess the Pharmacokinetics, Safety and Tolerability of Multiple Administrations of 30 mg PMI-150 (Intranasal Ketamine) in Healthy Adult Volunteers
Brief Title: Multiple Dose Pharmacokinetics of Intranasal Ketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Javelin Pharmaceuticals, Javelin Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: KET-PK-002
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2008-01

CONDITIONS: Healthy
Keywords: pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment A (Experimental): intranasal ketamine
  Interventions: Drug: intranasal ketamine

INTERVENTIONS:
Drug: intranasal ketamine — intranasal ketamine

SUMMARY:
This is an open label, single-center study of the pharmacokinetic and safety profile of repeat doses of PMI-150 (intranasal ketamine) 30 mg in healthy adult volunteers.

DETAILED DESCRIPTION:
To examine safety and characterize the repeat dosing plasma profile, effect on absorption, and accumulation following repeated administration of 30 mg doses of PMI-150 (intranasal ketamine) to healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | multiple

CONTACTS AND LOCATIONS:
Overall Officials: Javelin Pharmaceuticals, Study Director — Javelin Pharmaceuticals